CLINICAL TRIAL: NCT01654809
Title: Evaluation of Safety and Immunogenicity Among Different Age-groups Receiving Different Split Influenza Vaccines
Brief Title: Safety and Immunogenicity Study of Split Influenza Virus Vaccine in Different Age Groups
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BJCDPC-1
Record Dates: First submitted 2012-07-28; First posted 2012-08-01 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- evaluated vaccine (Experimental): 0.25 mL, Intramuscular (infant/children dose) 0.5 mL, Intramuscular (adult dose)
  Interventions: Biological: evaluated vaccine; Biological: imported compared vaccine; Biological: domestic compared vaccine
- imported compared vaccine (Active Comparator): 0.25 mL, Intramuscular (infant/children dose) 0.5 mL, Intramuscular (adult dose)
  Interventions: Biological: evaluated vaccine; Biological: imported compared vaccine; Biological: domestic compared vaccine
- domestic compared vaccine (Active Comparator): 0.25 mL, Intramuscular (infant/children dose) 0.5 mL, Intramuscular (adult dose)
  Interventions: Biological: evaluated vaccine; Biological: imported compared vaccine; Biological: domestic compared vaccine

INTERVENTIONS:
Biological: evaluated vaccine — 0.25 mL, Intramuscular (infant/children dose) 0.5 mL, Intramuscular (adult dose)
Biological: imported compared vaccine — 0.25 mL, Intramuscular (infant/children dose) 0.5 mL, Intramuscular (adult dose)
Biological: domestic compared vaccine — 0.25 mL, Intramuscular (infant/children dose) 0.5 mL, Intramuscular (adult dose)

SUMMARY:
The purpose of this study is to observe the adverse reaction ratio and hemagglutination inhibition (HI) antibody positive rate, Geometric mean titer (GMT) of three brands split influenza virus vaccine in different population.

DETAILED DESCRIPTION:
Observational Objectives:

To describe the safety of evaluated vaccine, given in the two-dose schedule in accordance with the Package Insert, in children aged ≥ 6 months to ≤ 36 months,6th to 12th birthday and ≥ 60th birthday.

To describe the immunogenicity of evaluated vaccine, given in the two-dose schedule in accordance with the Package Insert, in children aged ≥ 6 months to ≤ 36 months, 6th to 12th birthday and ≥ 60rd birthday.

ELIGIBILITY:
Inclusion Criteria:

* participants were enrolled (toddlers: 6 months to 3 years; school-aged children: 6 to 12 years and older adults: ≥60 years）
* Eligible participants were generally healthy or had stable chronic medical conditions (for older adults only)

Exclusion Criteria:

* History of allergic reaction to any component of the study vaccines or previous influenza vaccine
* History of systemic hypersensitivity to hens' eggs
* History of Guillain Barré syndrome following administration of any influenza vaccine
* Any immunodeficient or immunocompromised conditions
* Receipt of cytotoxic or immunosuppressive drugs within the past 6 months
* Receipt of blood-derived product within the past 3 months
* Receipt of any vaccine within one month prior to study entry with exception of paediatric routine vaccination
* Receipt of non-study 2010-2011 seasonal TIV
* Participation in any other study with a non-approved drug during the study
* Acute febrile disease and other self-limiting illness were the temporary exclusion criteria

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2010-08; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the immunogenicity of evaluated vaccine | 6 months
  The immunologic equivalence of 7days after vaccination of influenza virus vaccine was measured in terms of GMTs.
To evaluate the safety | 4 months
  The incidence of adverse events was analyzed statistically

CONTACTS AND LOCATIONS:
Overall Officials: Nianmin Shi, Master, Study Chair — Beijing Chaoyang District Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Sanhe Centre for Disease Control and Prevention, Langfang, Hebei
  - Jiuyuan Center for Disease Control and Prevention, Baotou, Inner Mongolia